CLINICAL TRIAL: NCT06661642
Title: Clinical Prediction of Post-surgical Pain: External Validation
Brief Title: Clinical Prediction of Post-surgical Pain
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Aalborg University Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Camilla Gaarsdal Uhrbrand, MD, PhD-fellow, Aarhus University Hospital
Other Study IDs: 23956082
Record Dates: First submitted 2024-10-25; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Acute Postoperative Pain; Chronic Post Operative Pain
Keywords: Acute postoperative pain; Chronic postoperative pain; Prediction; Risk tool
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgery patients: Patients undergoing various elective and sub-acute surgical procedures including thoracic, cardiac, abdominal, vascular, plastic, spinal neurosurgery, and orthopaedic procedures.

SUMMARY:
This study aims to externally validate two clinical prediction models for moderate-to-severe acute post-surgical pain and chronic post-surgical pain. This multi-centre, prospective cohort study will be conducted in Denmark and will include adult patients undergoing various types of elective or sub-acute surgical procedures.

DETAILED DESCRIPTION:
Based on sample size calculations for prediction model validation, a total of 482 patients are required validation of the acute post-surgical pain model and 748 (575 + 30% for loss to follow-up) patients are required for validation of the chronic post-surgical pain model. Therefore, we will aim to recruit 748 patients in total.

ELIGIBILITY:
Inclusion Criteria:

All patients ≥ 18 years undergoing elective or sub-acute surgery

Exclusion Criteria:

Cognitive impairment not allowing for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective or sub-acute surgery meeting inclusion and exclusion criteria, including thoracic, cardiac, abdominal, vascular, plastic, neurosurgery and orthopaedic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 748 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Moderate-to-severe acute post-surgical pain | First 3 postoperative hours or until discharge from the PACU
  Worst pain intensity score at rest ≥ 4 on an 11-point numeric rating scale (NRS; 0-10) in the post-anaesthesia care unit (PACU) following surgery, where 0=no pain and 10=worst pain imaginable.
Chronic post-surgical pain | 3 months post-surgery
  Pain related to the surgical procedure measured as average pain intensity on rest or movement ≥ 3 in the past one week using an 11-point numeric rating scale (NRS; 0-10) where 0=no pain and 10=worst pain imaginable and average pain interference ≥ 3 using 11-point NRS among any one of seven short-form Brief Pain Inventory items (general activity, mood, walking ability, normal work (including housework), relations with other people, sleep, enjoyment of life) in the past one week, where 0=pain does not interfere and 10=pain completely interferes.

SECONDARY OUTCOMES:
Severe acute post-surgical pain | First 3 postoperative hours or until discharge from the PACU
  Worst pain intensity score at rest ≥ 7 on an 11-point numeric rating scale (NRS; 0-10) in the post-anaesthesia care unit (PACU) following surgery, where 0=no pain and 10=worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Lone Nikolajsen, Principal Investigator — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Bispebjerg and Frederiksberg Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No